CLINICAL TRIAL: NCT00433758
Title: Evaluation of the Performance and Use of the GlucoTrack(TM), Non-Invasive Glucose Monitoring Device
Brief Title: Evaluation of the GlucoTrack, Non-Invasive Glucose Monitoring Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Integrity Applications Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IA-A2-2007-01-CTIL
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2007-09

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus; Gestational Diabetes
Keywords: Diabetes; Blood glucose monitoring; Non invasive Blood glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes, Gestational; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: GlucoTrack — GT

SUMMARY:
The purpose of this study is to demonstrate the performance of the GlucoTrack device (non invasive device) in measuring blood glucose levels

DETAILED DESCRIPTION:
Diabetes is a leading cause of death in the Western World with medical costs increasing annually. There is no cure for diabetes, and blood glucose monitoring is a key component in diabetes treatment and management. Consistently high blood sugar levels can, over time, lead to complications such as blindness, kidney disease, heart disease, and nerve damage.In addition, low blood sugars may lead to immediate dangers. Self-monitoring of blood glucose levels is essential to the self-management of diabetes and has become widespread over the past decade. Blood glucose determinations are currently done by invasive methods (finger tip pricking), followed by measuring the blood drop characteristics. Currently, there is no commercially available reliable non-invasive glucose measurement device that being marketed.

The GlucoTrack, non-invasive device for determining glucose levels based on the simultaneous measurement of three independent orthogonal parameters.

The rationale for development of the device is to improve the patient's quality of life by providing a device that is easily used and provides a painless measurement method, thereby leading to higher compliance, and to better managed diabetes

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1, Type 2, or Gestational Diabetes
* Above the age of 10

Exclusion Criteria:

* Does not meet inclusion criteria
* Patients requiring dialysis
* Participation in other clinical investigations within the previous month.
* Pregnancy(excluding patients that intend to participate in the gestational group)

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2006-12; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Clarke Error Grid | Clarke Error Grid

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Harman-Boehm, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel